CLINICAL TRIAL: NCT01307813
Title: Evaluation of a Novel Endoscopic Suturing Device in a Treat and Resect Model
Brief Title: Apollo Overstitch, a Treat and Resect Model
Acronym: Overstitch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey Marks, MD, General Surgeon, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-10-31
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Results first posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Colon Malignant Tumor; Colon Benign Tumor
Keywords: colon distal; surgical resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic suturing device (Experimental): Assess the safety and effectiveness of the Apollo endoscopic suturing device (Overstitch) and cinching device for placement of sutures and surgical knots in a segment of colon under laparoscopic or open visualization of the operative area.
  Interventions: Device: Overstitch Endoscopic Suturing System

INTERVENTIONS:
Device: Overstitch Endoscopic Suturing System — Assess the safety and effectiveness of the Apollo endoscopic suturing device (Overstitch) and cinching device for placement of sutures and surgical knots in a segment of colon under laparoscopic or open visualization of the operative area.
  Patients will already require resection of segments of colon for treatment of benign or malignant disease and this will therefore be a treat and resect model
  Other Names: Endoscopic suturing and cinching device; for placement of sutures and surgical knots

SUMMARY:
The Overstitch (Apollo Endosurgery, Austin, Texas) is an FDA cleared product which attaches to a standard double channel endoscope. The Overstitch can place sutures under endoscopic guidance, with the goal of reproducing standard surgical techniques. These would include hemostasis, tissue approximation, anastomosis formation, fixation of intraluminal devices, or repair/closure of mucosal or full thickness defects such as perforations or endoscopic mucosal resection (EMR) sites. Knot tying of the endoscopically placed sutures is provided by an endoscopic cinching device that passes through the channel of the endoscope.

This feasibility trial will evaluate the ability of the Apollo suturing device (Overstitch) to endoscopically place sutures into normal mucosa, and then "tie" the sutures with the cinching device. These devices have been utilized effectively in explant, live porcine, and human cadaver colon and stomach models. In this treat and resect model, sutures would be placed in a segment of colon or stomach that is being surgically removed via open or laparoscopic technique for the treatment of benign or malignant disease. The sutures would be placed in a segment of normal mucosa remote to the pathology being surgically treated. In addition, the sutures will be placed under direct observation via laparoscopic or open visualization. After resection of the segment of colon, it will be evaluated grossly for level of suture placement, evidence of perforation, and quality of suture approximation with the cinching device.

DETAILED DESCRIPTION:
During the colectomy procedure, the intended proximal and distal margins of resection will be determined, and the protocol will proceed only if it is fully determined that the tissue will be fully resectable. The overstitch device affixed to a standard double channel gastroscope will then be advanced transanally into the segment of planned resected colon, away from the area of disease so as to not interfere with oncologic principles or post-resection pathologic evaluation. Endoscopic sutures and knot tying cinching elements will be placed, with a limit of 15 minutes for the total procedure. The entire procedure will be closely monitored under laparoscopic or open surgical visualization. After suture placement, the surgical resection will continue as planned. The specimen will then be examined for depth of suture placement, evidence of perforation, and quality of the suture approximation with the knot tying element.

ELIGIBILITY:
Inclusion Criteria:

* The patient population in this study will be candidates of either sex, over 18' who have an established indication for a surgical procedure requiring resection of a portion of colon distal to the splenic flexure. This will include both benign and malignant diseases.

Exclusion Criteria:

* Any underlying pathology in the determination of investigator that subject cannot undergo scoping
* Sutures cannot be placed in segment of bowel that will be included in the surgical resection
* Pregnant women will be excluded from participating in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Marks, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Endoscopic Suturing Device: Assess the safety and effectiveness of the Apollo endoscopic suturing device (Overstitch) and cinching device for placement of sutures and surgical knots in a segment of colon under laparoscopic or open visualization of the operative area.
  Overstitch Endoscopic Suturing System: Assess the safety and effectiveness of the Apollo endoscopic suturing device (Overstitch) and cinching device for placement of sutures and surgical knots in a segment of colon under laparoscopic or open visualization of the operative area.
  Patients will already require resection of segments of colon for treatment of benign or malignant disease and this will therefore be a treat and resect model
Period: Overall Study
Arm/Group | Endoscopic Suturing Device
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endoscopic Suturing Device
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Successful Suture Approximation With Cinching Device
Description: Assess the safety and effectiveness of the Apollo endoscopic suturing device (Overstitch) and cinching device for placement of sutures and surgical knots in a segment of colon under laparoscopic or open visualization of the operative area.
  The quality of cinch element effectiveness was graded on a four-point Likert scale (1 = Poor, 2 = Good, 3 = Very Good, 4 = Excellent).
Time Frame: Approximately 1 hour post resection of the colon in surgery
Population: Participants who received Overstitch.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Endoscopic Suturing Device
Number analyzed (Participants) | 4
score on a scale | 3.57 (0.72)

2. Primary Outcome: Successful Suture Approximation With Cinching Device
Description: Assess the safety and effectiveness of the Apollo endoscopic suturing device (Overstitch) and cinching device for placement of sutures and surgical knots in a segment of colon under laparoscopic or open visualization of the operative area.
  When two tissue bites were taken within an individual stitch, the quality of mucosal approximation was graded on a four-point Likert scale (1 = Poor, 2 = Good, 3 = Very Good, 4 = Excellent).
Time Frame: Approximately 1 hour post resection of the colon in surgery
Population: Participants who received Overstitch when two tissue bites were taken within an individual stitch.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Endoscopic Suturing Device
Number analyzed (Participants) | 3
score on a scale | 2.66 (0.94)

ADVERSE EVENTS:
Time Frame: Adverse intra-operative and post-operative events approximately 1 hour post resection of the colon in surgery were noted.
Arm/Group | Endoscopic Suturing Device
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No